CLINICAL TRIAL: NCT02597907
Title: Postoperative Nausea and Vomiting: Ramosetron Plus Aprepitant vs Palonosetron Plus Aprepitant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KNUH 2014-05-016
Record Dates: First submitted 2015-10-31; First posted 2015-11-05 (Estimated); Results first posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant; Palonosetron; ramosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aprepitant plus palonosetron (Experimental): aprepitant 80 mg palonosetron 0.075 mg
  Interventions: Drug: aprepitant; Drug: palonosetron
- aprepitant plus ramosetron (Active Comparator): aprepitant 80 mg ramosetron 0.3 mg
  Interventions: Drug: aprepitant; Drug: Ramosetron

INTERVENTIONS:
Drug: aprepitant — aprepitant 80 mg is given to all patients before surgery
Drug: palonosetron — palonosetron 0.075 mg is given to patients in the aprepitant plus palonosetron group after induction of general anesthesia
  Arms: aprepitant plus palonosetron
Drug: Ramosetron — ramosetron 0.3 mg is given to patients in the aprepitant plus ramosetron group after induction of general anesthesia
  Arms: aprepitant plus ramosetron

SUMMARY:
The purpose of this study was to compare the antiemetic efficacy of aprepitant plus palonosetron versus aprepitant plus ramosetron in high risk patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
The purpose of this study was to compare the antiemetic efficacy of aprepitant plus palonosetron versus aprepitant plus ramosetron in high risk patients undergoing laparoscopic cholecystectomy.

Study is performed during 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non smoking, female patients, scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Patients with gastrointestinal disorder,
* Patients with allergies to any study medication,
* Patients who had received any sedatives, opioid, steroid or antiemetics within 24 h before surgery

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aprepitant Plus Ramosetron | Aprepitant Plus Palonosetron
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant Plus Palonosetron | Aprepitant Plus Ramosetron | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 44 | 88
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (10.6) | 48.8 (10.2) | 48.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Korea, Republic of | 44 | 44 | 88

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Postoperative Nausea and Vomiting
Description: The incidence of postoperative nausea and vomiting during 24 hours postoperatively
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Aprepitant Plus Palonosetron | Aprepitant Plus Ramosetron
Number analyzed (Participants) | 44 | 44
Participants | 5 | 18
Statistical Analysis 1: Comparison: Aprepitant Plus Palonosetron vs Aprepitant Plus Ramosetron; Test type: Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Aprepitant Plus Palonosetron | Aprepitant Plus Ramosetron
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes